CLINICAL TRIAL: NCT03949062
Title: A Phase 2, Open-Label Study to Evaluate the Safety and Efficacy of iR2 (Ibrutinib，Lenalidomide, Rituximab）in Untreated and Unfit Elderly Patients With Diffuse Large B-cell Lymphoma
Brief Title: Study Evaluating the Safety and Efficacy of iR2 in Untreated and Unfit Elderly Patients With DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director，Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL-iR2
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: iR2
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibrutinib; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iR2 (Experimental): Participants received six 21-day cycles of ibrutinib, lenalidomide, and rituximab (iR2) treatment (21-day cycles).
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 560mg per day administered orally on Day 1-21 of each 21-day cycle for 6 cycles
  Other Names: Imbruvica
Drug: Lenalidomide — Lenalidomide 25mg per day administered orally on Day 1-10 of each 21-day cycle for 6 cycles
  Other Names: Relvimid
Drug: Rituximab — Rituximab 375mg/m2 per day administered intraveneously on Day 1 of each 21-day cycle for 6 cycles
  Other Names: Rituxan

SUMMARY:
This is a single-arm, open-label phase 2 study of iR2 in the treatment of unfit and elderly patients with untreated diffuse large B-cell lymphoma。

DETAILED DESCRIPTION:
This open-label, single arm study will evaluate the efficacy and safety of ibrutinib， lenalidomide, rituximab (iR2) in previously untreated and unfit elderly subjects with diffuse large B-cell lymphoma. Subjects will receive 6 cycles of ibrutinib 560mg, day 1-21, orally (PO) , lenalidomide 25mg, day 1-10, rituximab 375mg/m2, intravenously, every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diffuse large B cell lymphoma, treatment naive
2. Age > 75 years
3. Ineligible for standard chemotherapy
4. Must has measurable lesion in CT or PET-CT prior to treatment
5. At least 3 months life expectation
6. Informed consented
7. No previous use of study drug

Exclusion Criteria:

1. Has accepted Chemotherapy before
2. Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
3. Lab at enrollment (Unless caused by lymphoma): Neutrophile<1.5*10^9/L ;Platelet<80*10^9/L; ALT or AST >2*ULN; AKP or bilirubin >1.5*ULN ;Creatinine>1.5*ULN
4. Not able to comply to the protocol for mental or other unknown reasons Pregnant or lactation
5. HIV infection
6. If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA,DNA positive patients cannot be enrolled.
7. Other uncontrollable medical condition that may that may interfere the participation of the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Overall response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with response(complete response and partial response) was determined on the basis of investigator assessments according to 2014 Lugano criteria
Progression free survival | Baseline up to data cut-off (up to approximately 4 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival in the overall study population was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Baseline up to data cut-off (up to approximately 4 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

OTHER OUTCOMES:
Circulating free Deoxyribonucleic Acid (cfDNA) monitoring | Baseline up to data cut-off (up to approximately 4 years)
  cfDNA in peripheral blood assessed by local lab

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, PhD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu PP, Shi ZY, Qian Y, Cheng S, Zhu Y, Jiang L, Li JF, Fang H, Huang HY, Yi HM, Ouyang BS, Wang L, Zhao WL. Ibrutinib, rituximab, and lenalidomide in unfit or frail patients aged 75 years or older with de novo diffuse large B-cell lymphoma: a phase 2, single-arm study. Lancet Healthy Longev. 2022 Jul;3(7):e481-e490. doi: 10.1016/S2666-7568(22)00123-4. PMID 36102758